CLINICAL TRIAL: NCT00597259
Title: Pegasys Plus Entecavir Versus Entecavir Alone for Hepatitis Be Antigen-Positive Chronic Hepatitis B
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Pei-Jer Chen, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200710028M; No other ID
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Chronic Hepatitis B
Keywords: hepatitis B, entecavir, pegylated interferon alfa-2a
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — peginterferon alfa-2a; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Pegasys plus Entecavir
- B (Active Comparator): Entecavir Alone
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Pegasys plus Entecavir — Pegasys 180 mcg in 0.5 mL solution administered sc once weekly for 24 weeks plus entecavir (0.5mg mg/capsule) 0.5 mg administered po daily for 24 weeks
  Arms: A
Drug: Entecavir — ETV 0.5 mg daily monotherapy for 144 weeks
  Arms: B

SUMMARY:
Although the best treatment choice for chronic hepatitis B is not clarified yet, certain therapeutic concepts could be derived from the experience of treating patients with chronic hepatitis C or human immunodeficiency virus (HIV) infection. A major advancement in treating hepatitis C or HIV infection has been the development of combination therapy. Whether the combination therapy using Peg-IFN alfa-2a plus ETV can achieve a long-term beneficial effect against ETV alone is not clarified. A prior single-arm pilot study suggested that similar combination therapy may be beneficial in patients with chronic hepatitis B. In this proposal, we thus hypothesize that the efficacy by using combination therapy with pegylated IFN alfa-2a plus ETV is superior to that by using ETV alone in that Peg-IFN may restore host immunity against HBV and prolonged ETV can maximize viral suppression.

The objective of this clinical trial is to evaluate the efficacy of the combination of Peg-IFN alfa-2a at a dose of 180 mcg administered subcutaneously per week and ETV 0.5 mg daily for 24 weeks followed by ETV 0.5 mg daily monotherapy for an additional 120 weeks versus ETV 0.5 mg daily monotherapy for 144 weeks in patients with HBeAg-positive chronic hepatitis B. It will be an open-label, randomized, comparative, multi-center clinical trial. The recruited patients will be equally randomized into two treatment groups. Treatment-free follow-up period will be 48 weeks in both groups of patients. All subjects will be assessed for loss of HBeAg, presence of anti-HBe, loss of HBsAg, presence of anti-HBs, suppression of HBV DNA, and normalization of serum ALT at the end of treatment and end of follow-up. Genotypic and virologic resistance to ETV will also be assessed at baseline and at end of years 1, 2 and 3. The primary efficacy will be HBeAg seroconversion.

DETAILED DESCRIPTION:
Currently, there are several antiviral treatments effective for suppression of viral replication but still failed to cure HBV infection in patients with chronic hepatitis B. The short-term treatment goals are thus to control hepatitis activity, to obtain hepatitis B e antigen (HBeAg) seroconversion, and to improve necroinflammatory activity and fibrosis of the liver. Six drugs have been worldwide approved for the treatment of chronic hepatitis B at present: conventional IFN (IFN) alfa, lamivudine (LAM), adefovir dipivoxil (ADV), pegylated IFN (Peg-IFN) alfa, entecavir (ETV) and recently telbivudine (LdT). Conventional IFN alfa monotherapy has a narrow range of efficacy, is associated with several adverse effects and is inconvenient because of frequent injections. Lamivudine is better tolerated; but virologic response to lamivudine is frequently not durable and prolonged lamivudine treatment is commonly associated with the emergence of drug-resistant HBV mutants. Adefovir dipivoxil is effective and has been approved for the treatment of chronic hepatitis B in many countries, but is nephrotoxic at doses higher than 10 mg per day for long time. Pegylated IFN alfa has been shown to be superior to conventional IFN alfa and lamivudine, and has already been approved for the treatment of chronic hepatitis B. Overall, satisfactory virologic and serologic responses could be achieved using pegylated IFN alfa alone in around 30-44% of these patients. Entecavir, a carbocyclic deoxyguanosine analog, which is active against both lamivudine- and adefovir dipivoxil-naïve and -resistant HBV, is the most potent anti-HBV agent ever discovered. In addition, the 4-year drug resistance rate is <1.0% in selected lamivudine-naïve patients. LdT is another thymidine nucleoside analogue with potent in vitro activity against HBV and approved for CHB. Recent phase III GLOBE trials have proved this agent to be more effective in the treatment of HBeAg+ve and -ve chronic hepatitis B than lamivudine. However, resistance to telbivudine was noted in around 10% of subjects after 104-week continuous therapy, although still fewer than that in patients receiving lamivudine.

Although the best treatment choice for chronic hepatitis B is not clarified yet, certain therapeutic concepts could be derived from the experience of treating patients with chronic hepatitis C or human immunodeficiency virus (HIV) infection. A major advancement in treating hepatitis C or HIV infection has been the development of combination therapy. Whether the combination therapy using Peg-IFN alfa-2a plus ETV can achieve a long-term beneficial effect against ETV alone is not clarified. A prior single-arm pilot study suggested that similar combination therapy may be beneficial in patients with chronic hepatitis B. In this proposal, we thus hypothesize that the efficacy by using combination therapy with pegylated IFN alfa-2a plus ETV is superior to that by using ETV alone in that Peg-IFN may restore host immunity against HBV and prolonged ETV can maximize viral suppression.

The objective of this clinical trial is to evaluate the efficacy of the combination of Peg-IFN alfa-2a at a dose of 180 mcg administered subcutaneously per week and ETV 0.5 mg daily for 24 weeks followed by ETV 0.5 mg daily monotherapy for an additional 120 weeks versus ETV 0.5 mg daily monotherapy for 144 weeks in patients with HBeAg-positive chronic hepatitis B. It will be an open-label, randomized, comparative, multi-center clinical trial. The recruited patients will be equally randomized into two treatment groups. Treatment-free follow-up period will be 48 weeks in both groups of patients. All subjects will be assessed for loss of HBeAg, presence of anti-HBe, loss of HBsAg, presence of anti-HBs, suppression of HBV DNA, and normalization of serum ALT at the end of treatment and end of follow-up. Genotypic and virologic resistance to ETV will also be assessed at baseline and at end of years 1, 2 and 3.

We anticipate the rate of HBeAg seroconversion, primary efficacy parameter, to be around 35% at the end of 3-year entecavir therapy, but decreases to be 30% at the end of 24-week post-treatment follow-up. We also anticipate that by combining Pegasys, the rate of seroconversion at the end of treatment is 50% and at the end of 24-week post-treatment follow-up could be 45%. With a 5% nominal significance level (one-sided), 128 patients per group under a 1:1 ratio (a total of 256 patients) will provide 80% power to detect a difference of 15% in treatment response rates between group I and II. Because this will be a 4-year study for each patient, we thus anticipate that the dropout rate may be as high as 15%. Accordingly, a total of 294 patients will be recruited, in order to account for a dropout rate of up to 15%.

A final analysis will be conducted when all patients have completed 144-week treatment and 48 weeks of follow-up. Primary and secondary efficacy parameters will be evaluated by an intention-to-treat analysis. Exact (1-sided) 95%-confidence interval from the binomial distribution will be provided for response rates in individual patient groups. All categorical and continuous variables will be analyzed by chi-square test and Student t test, respectively. For continuous variables with outliers, nonparametric test will be used instead. The analysis of histologic response will include only those who receive the pre- and post-treatment biopsy.

ELIGIBILITY:
Inclusion criteria:

Subjects meeting all of the following criteria will be considered for entering the study:

1. Adult male or female, 18 to 70 years of age

   * Patient must have documented positive serum HBsAg for a minimum of 6 months prior to entry into study.
   * Patients must show evidence of HBV replication and hepatitis documented by

     * Positive serum HBV DNA within 3 months prior to entry (HBV DNA >100,000 copies/mL)
     * Positive serum HBeAg within 3 months prior to entry.
     * Documented presence of abnormal alanine aminotransferase (ALT) twice within 3 months prior to entry (2 to 10 folds above the upper normal level)
     * Liver biopsy finding shows evidence of chronic hepatitis without liver cirrhosis
     * Naïve to lamivudine
2. Compensated liver disease with the following minimum hematological and serum biochemical criteria:

   * Hemoglobin values of ≥ 12 gm/dL for both genders
   * WBC ≥ 3,000/mm3
   * Neutrophil count ≥ 1,500/ mm3
   * Platelets ≥ 100,000/ mm3
   * PT prolong < 3 sec, INR < 1.2
   * Total bilirubin ≤ 2 mg/dL
   * Albumin > 3.5 g/dL
   * Uric acid within normal ranges
   * Serum creatinine ≤ 123.76 mmol/L (≤ 1.4 mg/dL)
   * Hemoglobin A1C ≤ 8.5% for diabetic patients (whether on medication and/or controlled with diet)
3. Thyroid stimulating hormone (TSH), within normal ranges (subjects requiring medication to maintain TSH levels in the normal range are eligible if all other inclusion/exclusion criteria are met)
4. Negative serum antibody to hepatitis C (anti-HCV)
5. Negative antibody to human immunodeficiency virus (anti-HIV)
6. Alfa-fetoprotein within normal range (obtained within the previous year, or if elevated and <100 ng/ml, then a negative ultrasound for hepatocellular carcinoma within prior 3 months is required.)
7. Subject must be willing to give written informed consent and be able to adhere to dose and visit schedules

Exclusion criteria:

Subjects presenting with any of the following will not be included in the study:

1. Women who are pregnant or nursing
2. Prior treatment for hepatitis with any interferon, NA or other investigational agents
3. Prior treatment for hepatitis with immunomodulatory drug within previous 2 years
4. Suspected hypersensitivity to interferon
5. Have evidence of cirrhosis
6. History of severe psychiatric disease, especially depression
7. Concurrent malignancies (including hepatocellular carcinoma)
8. Unstable or significant cardiovascular diseases (e.g., angina, congestive heart failure, recent myocardial infarction, severe hypertension or significant arrhythmia; subjects with ECG showing clinically significant abnormalities)
9. Prolonged exposure to known hepatotoxins such as alcohol or drugs
10. History of thyroid disease poorly controlled on prescribed medication
11. Poorly controlled diabetes mellitus
12. Have suspected or confirmed significant hepatic disease from an etiology other than HBV (e.g., alcohol, autoimmune disease etc.)
13. Patients co-infected with hepatitis C and /or HIV
14. Severe renal disease or myeloid dysfunction
15. History of organ transplantation other than cornea and hair transplant
16. Any medical condition requiring, or likely to require during the course of the study, chronic systemic administration of steroids
17. Any other condition which in the opinion of the investigator would make the subject unsuitable for enrollment, or could interfere with the subject participating in and completing the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2008-01; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
HBeAg seroconversion | at the end of 24 weeks post-treatment follow-up

SECONDARY OUTCOMES:
Serum ALT normalization, HBeAg loss, serum HBV DNA disappearance, HBsAg disappearance, histologic change, entecavir resistance | At the end of treatment and 24 weeks after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Jer Chen, M.D., Ph.D., Principal Investigator — National Taiwan University Hospital Department of Internal Medicine
Locations (1):
- National Taiwan University Hospital Department of Internal medicine, Taipei, Taiwan